CLINICAL TRIAL: NCT01262820
Title: A Multi-Center Open Label Phase II Study of Pazopanib in Stage IIIB/IV Non-Squamous Non-Small Cell Lung Cancer After Progression on First Line Therapy Containing Bevacizumab
Brief Title: Pazopanib In Stage IIIB/IV NSCLC Lung Cancer After Progression on First Line Therapy Containing Bevacizumab
Acronym: LCCC0921
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0921; NCT01107652 (obsolete NCT alias)
Record Dates: First submitted 2010-12-07; First posted 2010-12-17 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: Pazopanib; Non Squamous Non Small Cell Lung Cancer; After Progress on first line therapy; Using Bevacizumab
MeSH Terms: conditions — Lung Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Intervention (Experimental): Subjects will take Pazopanib, 800 mg daily by mouth throughout the time in study
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib, 800 mg by mouth daily each 21 day cycle

SUMMARY:
This is an open label Phase II Trial that using the investigational anti-cancer agent, Pazopanib to see whether non-squamous non-small cell lung cancer will respond to its use by decreasing the size of the tumor or stopping its growth.

DETAILED DESCRIPTION:
This multi-centered phase II trial will examine pazopanib stage IIIB/IV non-squamous NSCLC patients who have progressed on first-line therapy containing bevacizumab. Treatment should continue until disease progression, unacceptable toxicity, study withdrawal, or death. Patients who progress will be treated at the discretion of their physician. all patients who initiate treatment will be evaluated for disease control rate, which is the primary endpoint of this study.

The primary objective is to estimate the disease control rate of pazopanib alone in patients with stage IIIB/IV non-squamous NSCLC who progressed while on bevacizumab. Disease control rate id defined as complete (CR) + partial response (PR) + stable disease (SD) lasting greater than or equal to 12 weeks as defined by RECIST.

Secondary Objectives To estimate the combined response rate (CR + PR) of pazopanib according to RECIST To estimate the progression free survival (defined as time of enrollment until disease progression or death) and overall survival (defined as time of enrollment until death) of patients treated with pazopanib.

To evaluate the safety and tolerability of pazopanib using the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.0 To explore potential correlations between blood biomarkers and clinical response.

Pazopanib is dosed continuously throughout the study. Cycle lengths are identified as 21 days for purposes of the calendar.

The treatment dosage and administration for participating subjects will be, Pazopanib, 800 mg by mouth daily during a 21 day cycle until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Stage IIIB (with malignant pleural or pericardial effusion or supraclavicular lymph node involvement) or stage IV NSCLC
* Evidence of progression while on bevacizumab
* Patients treated for CNS metastases who are asymptomatic with no requirement for steroids for 2 weeks prior to first dose of study drug

Exclusion Criteria:

* Prior malignancy
* Clinically significant gastrointestinal abnormalities
* Presence of uncontrolled infection or nonhealing wound, fracture, or ulcer
* History of cardiovascular conditions within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stinchcombe, MD, Principal Investigator — North Carolina Cancer Hospital at University of NC at Chapel Hill
Locations (2):
- United States (2):
  - North Carolina Cancer Hospital at U of North Carolina at CH, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: web address for Lineberger Comprehensive Cancer Center at UNC — http://unclineberger.org
- See also: web address for the National Cancer Institute (NCI) — http://cancer.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between April 2010 and January 2014
Pre-assignment Details: A total of 22 patients provided informed consent for this trial; 7 patients were considered ineligible leaving 15 patients who enrolled and were treated on study.
Period: Overall Study
Arm/Group | Single Intervention
Started | 15
Completed | 0
Not Completed | 15
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 9
Not completed — Drug held for 21+ days | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Intervention
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Response (CR + PR + SD) as defined by RECIST v1.1 lasting equal to or greater than 12 weeks in patients treated with pazopanib alone for stage IIIB/IV non-squamous NSCLC after progression on first line therapy containing bevacizumab Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) : Complete Response (CR) is defined as Disappearance of all target lesions; Partial Response (PR), as a >=30% decrease in the sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) of all target lesions; Progression, as a 20% increase in the sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) of all target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. Target lesions are representative of all involved organs and measurable by radiographic imaging.
Time Frame: Eight (8) months w additional time for response date to mature (up to 2 years per participant)
Measure: Number (95% Confidence Interval); unit: % of participants with disease control
Arm/Group | Single Intervention
Number analyzed (Participants) | 15
% of participants with disease control | 13 [2 to 40]

2. Secondary Outcome: Combined Response Rate (CR + PR) of Pazopanib According to RECIST v1.1
Description: Estimate of combined response rate (Complete Response (CR) + Partial Response (PR) per RECIST v1.1 Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) : Complete Response (CR) is defined as the disappearance of all target lesions and Partial Response (PR) as a >=30% decrease in the sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) of all target lesions.Target lesions are representative of all involved organs and measurable by radiographic imaging.
Time Frame: 8 months with additional time for response to mature (up to 2 years per participant)
Measure: Number; unit: participants
Arm/Group | Single Intervention
Number analyzed (Participants) | 15
participants | 0

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as time of enrollment until disease progression or death Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) : Progression is defined as a 20% increase in the sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) of all target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Target lesions are representative of all involved organs and measurable by radiographic imaging.
Time Frame: Eight (8) months w additional time for response data to mature (up to 2 years per participant)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Single Intervention
Number analyzed (Participants) | 15
weeks | 10.9 [8.1 to 18.9]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time of enrollment until death
Time Frame: Eight (8) months w additional time for response date to mature (up to 2 years per participant)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Single Intervention
Number analyzed (Participants) | 15
weeks | 24.1 [20.3 to 33.7]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Single Intervention
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Intervention (N=15)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Lung Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pericardial Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) — due to lung cancer
Vomiting (Gastrointestinal disorders) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) — due to metastatic disease
intracranial hemorrhage (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — bile duct obstruction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Intervention (N=15)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 3 (6)
Alkaline Phosphatase Increased (Investigations) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 9 (9)
Anxiety (Psychiatric disorders) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 5 (8)
Blood Bilirubin Increased (Investigations) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Esophageal Pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (12)
Fever (General disorders) | 1 (4)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Ggt Increased (Investigations) | 2 (5)
Headache (Nervous system disorders) | 1 (4)
Hemoglobin Increased (Investigations) | 1 (1)
Hepatitis viral (Hepatobiliary disorders) | 1 (1)
Hot Flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Lipase Increased (Investigations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 2 (2)
Mucositis Oral (Gastrointestinal disorders) | 3 (7)
Nausea (Gastrointestinal disorders) | 8 (14)
Neutrophil Count Decreased (Investigations) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Oral Hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (3)
Platelet Count Decreased (Investigations) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Pruitus (Skin and subcutaneous tissue disorders) | 1 (1)
Renal And Urinary Disorders - Other, Specify (Renal and urinary disorders) | 1 (1) — Dyduria
Skin And Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (3) — Hair color changes (white at scalp)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (10)
Weight Loss (Investigations) | 5 (5)
White Blood Cell Decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes